CLINICAL TRIAL: NCT03285477
Title: A Phase 3, Double-Blind, Vehicle-Controlled, Randomized, Parallel Group, Multicenter, Efficacy and Safety Study of KX2-391 Ointment 1% in Adult Subjects With Actinic Keratosis on the Face or Scalp
Brief Title: A Multi-Center Study to Evaluate the Efficacy and Safety of KX2-391 Ointment 1% on AK on Face or Scalp
Acronym: AK003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KX01-AK-003; U1111-1191-8233 (Other: UTN)
Record Dates: First submitted 2017-09-07; First posted 2017-09-18 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratosis; Keratosis; Keratosis, Actinic; Skin Diseases; Actinic Keratoses; Precancerous Conditions; Neoplasms
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Skin Diseases; Precancerous Conditions; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study tested KX2-391 Ointment 1% against a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Central Vendors and the sponsor were masked. The sponsor was unblind at the end of Day 57.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Vehicle Ointment was applied topically once daily for 5 consecutive days on face or scalp
  Interventions: Drug: Placebo
- KX2-391 Ointment 1% (Experimental): KX2-391 Ointment 1% was applied topically once daily for 5 consecutive days on face or scalp
  Interventions: Drug: KX2-391 Ointment 1%

INTERVENTIONS:
Drug: Placebo — Vehicle Ointment was used in participants with Clinically typical AK on the face or scalp.
  Arms: Placebo
Drug: KX2-391 Ointment 1% — The experimental drug, KX2-391 Ointment 1% was used in participants with Clinically typical AK on the face or scalp.
  Arms: KX2-391 Ointment 1%

SUMMARY:
This Phase III study is designed to evaluate the efficacy and safety of KX2-391 Ointment in adult participants when applied to an area of skin containing 4-8 stable, clinically typical Actinic Keratosis (AK) lesions on the face or scalp.

DETAILED DESCRIPTION:
This study was a double-blinded, multicenter, activity, and safety study of KX2-391 Ointment administered topically to the face or scalp of participants with actinic keratosis.

The study consists of Screening, Treatment, Follow-up, and Recurrence Follow-up Periods. Eligible participants received 5 consecutive days of topical treatment, to be applied at the study site. Activity (lesion counts) and safety evaluations was performed.

ELIGIBILITY:
Inclusion Criteria

1. Males and females greater than or equal to (≥) 18 years old
2. A defined area on the face or scalp contains 4 to 8 clinically typical, visible, and discrete AK lesions
3. Participants who in the judgment of the Investigator, are in good general health
4. Females must be postmenopausal [greater than (>) 45 years of age with at least 12 months of amenorrhea], surgically sterile (by hysterectomy, bilateral oophorectomy, or tubal ligation); or, if of childbearing potential, must be using highly effective contraception for at least 30 days or 1 menstrual cycle, whichever is longer, prior to study treatment and must agree to continue to use highly effective contraception for at least 30 days following their last dose of study treatment. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive implant, injection or patch, intrauterine device or complete abstinence from sexual intercourse.
5. Sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to use barrier contraception from Screening through 90 days after their last dose of study treatment.
6. All participants must agree not to donate sperm or eggs or attempt conception from Screening through 90 days following their last dose of study treatment
7. Willing to avoid excessive sun or UV exposure
8. Able to comprehend and are willing to sign the informed consent form (ICF).

Exclusion Criteria

1. Clinically atypical and/or rapidly changing AK lesions on the treatment area
2. Location of the selected area is:

   * On any location other than the face or scalp
   * Within 5 cm of an incompletely healed wound
   * Within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
3. Been previously treated with KX2-391 Ointment
4. Anticipated need for in-patient hospitalization or in-patient surgery from Day 1 to Day 57
5. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within the treatment area or within 2 cm of the treatment area, within 8 weeks prior to the Screening visit
6. Use of the following therapies and/or medications within 2 weeks prior to the Screening visit:

   * Cosmetic or therapeutic procedures (eg, use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treatment area
   * Acid-containing therapeutic products (eg, salicylic acid or fruit acids, such as alpha- and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treatment area
   * Topical salves (non-medicated/non-irritant lotion and cream are acceptable) or topical steroids within the treatment area or within 2 cm of the selected treatment area; artificial tanners within the treatment area or within 5 cm of the selected treatment area
7. Use of the following therapies and/or medications within 4 weeks prior to the Screening visit:

   * Treatment with immunomodulators (eg, azathioprine), cytotoxic drugs (eg, cyclophosphamide, vinblastine, chlorambucil, methotrexate) or interferons/interferon inducers
   * Treatment with systemic medications that suppress the immune system (eg, cyclosporine, prednisone, methotrexate, alefacept, infliximab)
8. Use of systemic retinoids (eg, isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit
9. A history of sensitivity and/or allergy to any of the ingredients in the study medication
10. A skin disease (eg, atopic dermatitis, psoriasis, eczema) or condition (eg, scarring, open wounds) that, in the opinion of the Investigator, might interfere with the study conduct or evaluations, or which exposes the participants to unacceptable risk by study participation
11. Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would expose the participant to unacceptable risk by study participation
12. Females who are pregnant or nursing
13. Participated in an investigational drug trial during which an investigational study medication was administered within 30 days or 5 half-lives of the investigational product, whichever is longer, before dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Fang, MD, Study Chair — Athenex, Inc.
Locations (30):
- United States (30):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Center For Dermatology Clinical Research, Fremont, California
  - Contour Dermatology, Rancho Mirage, California
  - Western States Clincial Research, Inc., Wheat Ridge, Colorado
  - Skin care Research, Inc, Boca Raton, Florida
  - Olympian Clinical Research, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Arlington Dermatology, Arlington Heights, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - DelRicht Research, New Orleans, Louisiana
  - ActivMed Practices & Research, Inc., Beverly, Massachusetts
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists PC, Omaha, Nebraska
  - JDR Dermatology Research, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai Beth Israel, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - PMG Research of Cary, Cary, North Carolina
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - PMG Research of Winston-Salem,LLC, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Synexus US, Greer, South Carolina
  - J&S Studies, Inc., College Station, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blauvelt A, Kempers S, Lain E, Schlesinger T, Tyring S, Forman S, Ablon G, Martin G, Wang H, Cutler DL, Fang J, Kwan MR; Phase 3 Tirbanibulin for Actinic Keratosis Group. Phase 3 Trials of Tirbanibulin Ointment for Actinic Keratosis. N Engl J Med. 2021 Feb 11;384(6):512-520. doi: 10.1056/NEJMoa2024040. PMID 33567191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 31 sites in United States from 18 September 2017 to 24 April 2019.
Pre-assignment Details: A total of 351 participants were enrolled in the study, 176 participants were randomized to the Vehicle control (121 face, 55 scalp treatment) and 175 participants were randomized to KX2-391 Ointment 1 percent (%) (119 face, 56 scalp treatment).
Period: Treatment and Response Assessment Period
Arm/Group | Placebo | KX2-391 Ointment 1%
Started | 176 | 175
Completed | 174 | 175
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawn of Consent | 1 | 0
Period: Recurrence Follow-up Period
Arm/Group | Placebo | KX2-391 Ointment 1%
Started (Number of participants who achieved 100% AK clearance at Day 57 visit and entered the recurrence follow-up period.) | 8 | 77
Completed | 2 | 22
Not Completed | 6 | 55
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal of consent | 1 | 3
Not completed — AK recurrence during the Recurrence Follow-Up Period | 5 | 51

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | KX2-391 Ointment 1% | Total
Number analyzed (Participants) | 176 | 175 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.41) | 69.5 (8.55) | 69.9 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 154 | 147 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 171 | 173 | 344
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 175 | 175 | 350
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of AK Lesions [Mean (Standard Deviation); unit: Lesions] | 5.9 (1.35) | 5.8 (1.28) | 5.8 (1.31)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete (100%) Clearance of Actinic Keratosis (AK) Lesions
Description: Complete clearance rate was defined as the percentage of participants at Day 57 with no clinically visible AK lesions in the treatment area.
Time Frame: Day 57
Population: ITT population included all participants randomized in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
percentage of participants | 5 | 44
Statistical Analysis 1: Comparison: Placebo vs KX2-391 Ointment 1%; Statistical significance in the study for Day 57 complete clearance rate was analyzed using a Cochran-Mantel-Haenszel model controlling for treatment location (face or scalp) and treatment group (Placebo versus KX2-391 Ointment 1%); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value threshold for statistical significance was 0.5%

2. Secondary Outcome: Percentage of Participants With Partial Clearance Rate of Actinic Keratosis Lesions at Day 57
Description: Partial clearance rate of AK lesions was defined as the percentage of participants with a greater than or equal to (>=) 75% reduction in the number of AK lesions identified at Baseline (Day 1 predose) in the treatment area.
Time Frame: Day 57
Population: ITT population included all participants randomized in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
percentage of participants | 16 | 68
Statistical Analysis 1: Comparison: Placebo vs KX2-391 Ointment 1%; Statistical significance in the study for Day 57 partial clearance rate was analyzed using a Cochran-Mantel-Haenszel model controlling for treatment location (face or scalp) and treatment group (Placebo versus KX2-391 Ointment 1%); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value threshold for statistical significance was 0.5%

3. Secondary Outcome: Overall Change From Baseline in Actinic Keratosis Lesion Counts at Days 8, 15, 29 and 57
Description: Overall the change from baseline in lesion count at each visit were summarized and reported using descriptive statistics by treatment location (face or scalp).
Time Frame: Days 8, 15, 29 and 57
Population: ITT population included all participants randomized in the study.
Measure: Median (Full Range); unit: lesion count
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
lesion count
  Day 8: number analyzed (Participants) | 172 | 135
  Day 8 | 0.0 [-7 to 3] | -1.0 [-8 to 4]
  Day 15: number analyzed (Participants) | 175 | 162
  Day 15 | 0.0 [-7 to 2] | -4.0 [-8 to 4]
  Day 29: number analyzed (Participants) | 173 | 174
  Day 29 | -1.0 [-7 to 4] | -4 [-8 to 1]
  Day 57: number analyzed (Participants) | 174 | 175
  Day 57 | -1.0 [-7 to 5] | -5.0 [-8 to 0]

4. Secondary Outcome: Percentage of Participants With Recurrence of Actinic Keratosis Lesions Who Achieved Complete Clearance at Day 57
Description: Recurrence rate was estimated based on Kaplan-Meier method, with recurrence define as appearance of any AK lesions in the treatment area, including those recurred or newly identified.
Time Frame: 3, 6, 9 and 12 months post-Day 57
Population: Recurrence Follow-up Population includes participants achieved complete clearance at the Day 57visit. The recurrence rate was evaluated only for KX2-391 Ointment 1% arm, pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | KX2-391 Ointment 1%
Number analyzed (Participants) | 77
percentage of participants
  3 Months Post-Day 57: number analyzed (Participants) | 76
  3 Months Post-Day 57 | 33
  6 Months Post-Day 57: number analyzed (Participants) | 50
  6 Months Post-Day 57 | 30
  9 Months Post-Day 57: number analyzed (Participants) | 33
  9 Months Post-Day 57 | 33
  12 months Post-Day 57: number analyzed (Participants) | 22
  12 months Post-Day 57 | 18

5. Secondary Outcome: Number of Participants With Maximal Post Baseline Local Skin Reaction (LSR)
Description: Maximal post baseline LSR was defined as the highest grade of any LSR reported at any post baseline visits for a participant. The LSR assessment was an Investigator's (or sub-investigator's) assessment of the following signs on the treatment area: erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration. The LSRs were graded on a 4-point scale ranging from 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense).
Time Frame: Day 57
Population: Safety analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants
  Erythema-Grade 0 | 81 | 6
  Erythema-Grade 1 | 84 | 48
  Erythema-Grade 2 | 11 | 116
  Erythema-Grade 3 | 0 | 5
  Flaking/Scaling-Grade 0 | 72 | 16
  Flaking/Scaling-Grade 1 | 90 | 70
  Flaking/Scaling-Grade 2 | 14 | 78
  Flaking/Scaling-Grade 3 | 0 | 11
  Crusting-Grade 0 | 140 | 84
  Crusting-Grade 1 | 33 | 69
  Crusting-Grade 2 | 3 | 20
  Crusting-Grade 3 | 0 | 2
  Swelling-Grade 0 | 163 | 107
  Swelling-Grade 1 | 12 | 55
  Swelling-Grade 2 | 1 | 12
  Swelling-Grade 3 | 0 | 1
  Vesiculation/Pustulation-Grade 0 | 174 | 158
  Vesiculation/Pustulation-Grade 1 | 2 | 14
  Vesiculation/Pustulation-Grade 2 | 0 | 2
  Vesiculation/Pustulation-Grade 3 | 0 | 1
  Erosion/Ulceration-Grade 0 | 168 | 155
  Erosion/Ulceration-Grade 1 | 8 | 15
  Erosion/Ulceration-Grade 2 | 0 | 5
  Erosion/Ulceration-Grade 3 | 0 | 0

6. Secondary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area
Description: Absence or presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment area were assessed.
Time Frame: Baseline (Day 1 predose), Days 5, 8, 15, 29 and 57
Population: Safety analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants
  Hypopigmentation: Baseline | 21 | 21
  Hypopigmentation: Day 5 | 19 | 11
  Hypopigmentation: Day 8 | 21 | 10
  Hypopigmentation: Day 15 | 23 | 12
  Hypopigmentation: Day 29 | 23 | 17
  Hypopigmentation: 57 | 20 | 13
  Hyperpigmentation: Baseline | 27 | 22
  Hyperpigmentation: Day 5 | 24 | 18
  Hyperpigmentation: Day 8 | 23 | 17
  Hyperpigmentation: Day 15 | 26 | 20
  Hyperpigmentation: Day 29 | 25 | 18
  Hyperpigmentation: Day 57 | 23 | 12
  Scarring: Baseline | 10 | 12
  Scarring: Day 5 | 8 | 8
  Scarring: Day 8 | 9 | 7
  Scarring: Day 15 | 7 | 8
  Scarring: Day 29 | 7 | 9
  Scarring: Day 57 | 7 | 7

7. Secondary Outcome: Number of Participants With Adverse Event (AE), Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Events of Special Interests
Description: An AE was defined as any untoward medical occurrence in participant which does not necessarily have causal relationship with treatment. An AE was any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal product, whether or not considered related to medicinal product. An SAE was any untoward medical occurrence that at any dose resulted in death; was life threatening; required persistent/significant disability/incapacity; resulted in initial or prolonged in patient hospitalization; was congenital anomaly/birth defect or otherwise considered medically important. TEAEs (serious and non-serious) were defined as either those AEs with onset after first dose or those pre-existing AEs that worsen after first dose. Events of special interest included skin cancers (including basal cell carcinoma, squamous cell carcinoma, melanoma and their location and treatment area), ocular exposure, overdose, and pregnancy.
Time Frame: Baseline (Day 1 predose) up to Day 57
Population: Safety analysis population included all randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants
  Participants with AE | 62 | 66
  Participants with any TEAE | 57 | 57
  Participants with SAE | 2 | 0
  Participants with events of special interest | 4 | 5

8. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, Events of Special Interests Within the Treatment Area After Day 57 and up to 12 Months Post-Day 57
Description: An AE was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. An SAE was any untoward medical occurrence that at any dose resulted in death; was life threatening; required persistent/significant disability/incapacity; resulted in initial or prolonged in patient hospitalization; was congenital anomaly/birth defect or otherwise considered medically important. Events of special interest included skin cancers (including basal cell carcinoma, squamous cell carcinoma, melanoma and their location and treatment area), ocular exposure, overdose, and pregnancy.
Time Frame: From Day 57 up to 12-months post-Day 57
Population: Recurrence Follow-up Population includes participants achieved complete clearance at the Day 57 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 8 | 77
Participants
  Participants with any AE | 0 | 4
  Participants with any SAE | 0 | 1
  Participants with events of special interest | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Hematology, Blood Chemistry, Urinalysis
Description: Assessed laboratory parameters included hematology, blood chemistry and urinalysis. Clinical significance and abnormal observations were determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants
  Hematology | 0 | 0
  Blood chemistry | 1 | 1
  Urinalysis | 0 | 3

10. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Vital Signs
Description: Vital signs included measurement of pulse rate, systolic and diastolic blood pressure, respiratory rate, and body temperature. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Physical Examination
Description: A physical examination included weight and height measurements was performed. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety analysis population included all randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Electrocardiograms (ECGs)
Description: ECG parameters included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 176 | 175
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1 predose) up to 15 months (12 months post-Day 57)
Description: Safety analysis population included all randomized participants who received at least one dose of study treatment.
Groups:
- Placebo: The Vehicle Ointment was applied topically once daily for 5 consecutive days on face or scalp
Arm/Group | Placebo | KX2-391 Ointment 1%
All-Cause Mortality (participants affected / at risk) | 1/176 | 0/175
Serious Adverse Events (participants affected / at risk) | 2/176 | 1/175
Other Adverse Events (participants affected / at risk) | 62/176 | 68/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | KX2-391 Ointment 1% (N=175)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | KX2-391 Ointment 1% (N=175)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Benign familial pemphigus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site discomfort (General disorders) | 0 (0) | 1 (1)
Application site dryness (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 6 (6) | 11 (23)
Application site paraesthesia (General disorders) | 1 (1) | 2 (2)
Application site pruritus (General disorders) | 8 (9) | 13 (14)
Application site warmth (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (3)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Protein urine (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (6)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-02-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03285477/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT03285477/SAP_001.pdf